CLINICAL TRIAL: NCT01784614
Title: Pharmacodynamics and Pharmacokinetics of Single Doses of LY2624803 in a 5-hour Phase Advance Model of Transient Insomnia in Healthy Japanese Subjects
Brief Title: A Study of LY2624803 in Japanese Participants With Transient Insomnia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 12662; I2K-JE-ZZAW (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-12

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 0.1 milligrams (mg) LY2624803 (Experimental): Single dose of 0.1 mg LY2624803 administered orally in up to 2 of 4 treatment periods
  Interventions: Drug: LY2624803 - Solution; Drug: Placebo - Capsule
- 1.0 mg LY2624803 (Experimental): Single dose of 1.0 mg LY2624803 administered orally in up to 2 of 4 treatment periods
  Interventions: Drug: LY2624803 - Capsule; Drug: Placebo - Solution
- 3.0 mg LY2624803 (Experimental): Single dose of 3.0 mg LY2624803 administered orally in up to 2 of 4 treatment periods
  Interventions: Drug: LY2624803 - Capsule; Drug: Placebo - Solution
- 6.0 mg LY2624803 (Experimental): Single dose of 6.0 mg LY2624803 administered orally in up to 2 of 4 treatment periods
  Interventions: Drug: LY2624803 - Capsule; Drug: Placebo - Solution
- Placebo (Placebo Comparator): Single dose of placebo administered orally in up to 1 of 4 treatment periods
  Interventions: Drug: Placebo - Solution; Drug: Placebo - Capsule

INTERVENTIONS:
Drug: LY2624803 - Solution — Administered orally as reconstituted solution
  Arms: 0.1 milligrams (mg) LY2624803
Drug: LY2624803 - Capsule — Administered orally as a capsule
  Arms: 1.0 mg LY2624803; 3.0 mg LY2624803; 6.0 mg LY2624803
Drug: Placebo - Solution — Administered orally as solution
  Arms: 1.0 mg LY2624803; 3.0 mg LY2624803; 6.0 mg LY2624803; Placebo
Drug: Placebo - Capsule — Administered orally as a capsule
  Arms: 0.1 milligrams (mg) LY2624803; Placebo

SUMMARY:
The aim of this study is to learn how different doses of LY2624803 affect sleep in healthy Japanese participants. The study has four treatment periods. Participants will receive a single dose of LY2624803 or placebo in each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or female Japanese
* Women of child-bearing potential, who test negative for pregnancy at the time of enrollment based on a urine pregnancy test and agree to use a reliable method of birth control during the study and for 3 months following the last dose of study drug
* Body mass index (BMI) of 17.6 to 26.4 kilogram per meter square (kg/m^2), inclusive
* Normal bedtime hours, with routine time spent in bed between 6.5 hours and 9 hours each night
* Clinical laboratory test results within normal reference range
* Venous access sufficient to allow blood sampling as per the protocol
* Are reliable and willing to make themselves available for the duration of the study and are willing and able to follow study procedures
* Have given written informed consent approved by Lilly and the ethical review board governing the site

Exclusion Criteria:

* Within 4 months of the initial dose of study drug, have received treatment with a drug that has not received regulatory approval for any indication
* Persons who have previously completed or withdrawn from this study or any other study investigating LY2624803 after receiving study drug
* Known allergies to LY2624803 or related compounds
* Women who are lactating
* Shift workers [those who shifted or plan to shift work within 7 days of any phase advance polysomnography (PSG) night] or any person who has crossed (or will have crossed) more than one time zone by aircraft within 3 days prior to entry
* Have an irregular or altered sleep/wake schedule that is likely to prevent from keeping a regular sleep/wake schedule during the study
* Regular napping (≥ 2 daytime naps/week by history)
* Extreme morning type or evening type
* Rhinitis, conjunctivitis, urticaria or chronic pain severe enough to interfere with sleep
* Nocturia that would interfere with sleep assessment
* Symptoms consistent with a sleep disorder or history of same
* Evidence of significant active neuropsychiatric disease and in particular evidence of significant medical or psychiatric illness within the past 12 months that could contribute to insomnia
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, neurocardiogenic or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* History or presence of orthostatic signs and symptoms within 2 years
* History of seizure or a close relative having a seizure disorder (such as epilepsy). History of a single febrile convulsion more than 10 years ago is acceptable. History of cranial trauma and loss of consciousness will be discussed prior to including any such participant
* Abnormal movements observed outside of normal sleep time
* Abnormal supine blood pressure and/or pulse rate
* Participants with orthostatic hypotension at screening
* An abnormality in the 12-lead electrocardiogram (ECG) that increases the risks associated with participating in the study
* Regular use of known drugs of abuse and/or positive findings on urinary drug screening
* Evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies
* Evidence of hepatitis C and/or positive hepatitis C antibody
* Evidence of hepatitis B and/or positive hepatitis B surface antigen
* Evidence of syphilis infection and/or positive syphilis test
* Use or intended use of prescription (except oral contraceptives), over-the-counter or herbal medication, specifically antihistamines, anticholinergic medications or any medications that affect sleepiness, within 28 days prior to Period 1 dosing and/or during the study
* Participants who have donated more than 200 milliliters (mL) of blood or component blood within one month of screening, or those who have donated more than 400 mL of blood within 3 months of screening
* History of smoking within the previous 6 months of screening
* Participants who have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), or participants unwilling to stop alcohol consumption for the period
* Participants whose daily caffeine intake does not permit maintenance of usual sleep/wake schedule
* No response to phase advance or a placebo responder
* Sleep disorders detected during the PSG screening night
* History or presence of breast cancer

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sagamihara, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a double-blind, randomized, placebo-controlled, 4-period cross-over study. The first 3 of which were used for polysomnography (PSG) measurements, and the fourth period was used to determine plasma concentrations of LY2624803 to estimate pharmacokinetic (PK) parameters.
Groups:
- Cohort 1: Period 1: Single dose of 1 placebo capsule plus placebo solution administered orally.
  Period 2: Single dose of one 1.0 milligram (mg) LY2624803 capsule plus placebo solution administered orally.
  Period 3: Single dose of one 3.0 mg LY2624803 capsule plus placebo solution administered orally.
  Period 4: Single dose of one 3.0 mg LY2624803 capsule plus placebo solution administered orally.
  There was at least 7 days washout between each period.
- Cohort 2: Period 1: Single dose of one 1.0 mg LY2624803 capsule plus placebo solution administered orally.
  Period 2: Single dose of 1 placebo capsule plus placebo solution administered orally.
  Period 3: Single dose of one 6.0 mg LY2624803 capsule plus placebo solution administered orally.
  Period 4: Single dose of one 6.0 mg LY2624803 capsule plus placebo solution administered orally.
  There was at least 7 days washout between each period.
- Cohort 3: Period 1: Single dose of one 3.0 mg LY2624803 capsule plus placebo solution administered orally.
  Period 2: Single dose of one 6.0 mg LY2624803 capsule plus placebo solution administered orally.
  Period 3: Single dose of 1 placebo capsule plus placebo solution administered orally.
  Period 4: Single dose of one 6.0 mg LY2624803 capsule plus placebo solution administered orally.
  There was at least 7 days washout between each period.
- Cohort 4: Period 1: Single dose of one 6.0 mg LY2624803 capsule plus placebo solution administered orally.
  Period 2: Single dose of one 3.0 mg LY2624803 capsule plus placebo solution administered orally.
  Period 3: Single dose of one 1.0 mg LY2624803 capsule plus placebo solution administered orally.
  Period 4: Single dose of one 1.0 mg LY2624803 capsule plus placebo solution administered orally.
  There was at least 7 days washout between each period.
- Cohort 5: Period 1: Single dose of 1 placebo capsule plus placebo solution administered orally.
  Period 2: Single dose of one 1.0 mg LY2624803 capsule plus placebo solution administered orally.
  Period 3: Single dose of one 3.0 mg LY2624803 capsule plus placebo solution administered orally.
  Period 4: Single dose of one 3.0 mg LY2624803 capsule plus placebo solution administered orally.
  There was at least 7 days washout between each period.
- Cohort 6: Period 1: Single dose of one 1.0 mg LY2624803 capsule plus placebo solution administered orally.
  Period 2: Single dose of 1 placebo capsule plus placebo solution administered orally.
  Period 3: Single dose of 0.1 mg LY2624803 solution plus 1 placebo capsule administered orally.
  Period 4: Single dose of 0.1 mg LY2624803 solution plus 1 placebo capsule administered orally.
  There was at least 7 days washout between each period.
- Cohort 7: Period 1: Single dose of one 3.0 mg LY2624803 capsule plus placebo solution administered orally.
  Period 2: Single dose of 0.1 mg LY2624803 solution plus 1 placebo capsule administered orally.
  Period 3: Single dose of 1 placebo capsule plus placebo solution administered orally.
  Period 4: Single dose of 0.1 mg LY2624803 solution plus 1 placebo capsule administered orally.
  There was at least 7 days washout between each period.
- Cohort 8: Period 1: Single dose of 0.1 mg LY2624803 solution plus 1 placebo capsule administered orally.
  Period 2: Single dose of one 3.0 mg LY2624803 capsule plus placebo solution administered orally.
  Period 3: Single dose of one 1.0 mg LY2624803 capsule plus placebo solution administered orally.
  Period 4: Single dose of 1.0 mg LY2624803 solution plus 1 placebo capsule administered orally.
  There was at least 7 days washout between each period.
Period: Period 1
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Received at Least 1 Dose of Study Drug | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 (One participant withdrew consent after completed Period 1 and did not enter Period 2.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2
Completed | 3 | 3 (One participant withdrew consent after completed Period 2 and did not enter Period 3.) | 3 | 3 | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Started | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2
Completed | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8
Started | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2
Completed | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Overall: Single dose of 0.1 mg LY2624803 oral solution plus 1 placebo capsule, one 1.0, 3.0 or 6.0 mg LY2624803 capsule plus placebo solution administered orally in up to 2 of 4 periods or 1 placebo capsule plus placebo solution administered orally in up to 1 of 4 periods.
  There was at least 7 days washout between each period.
Arm/Group | Overall
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 24

OUTCOME MEASURES:

1. Primary Outcome: Wake After Sleep Onset (WASO) With LY2624803 Compared to Placebo
Description: WASO was calculated as total time in awake epochs between sleep onset time (first stage 2 epoch) and the end of the primary recording period (8 hours after lights -off). Data presented are Geometric Least Squares (LS) means. Geometric LS mean was calculated using mixed models analysis. The model included factors for treatment, treatment sequence, period and participants.
Time Frame: 8 hours in Periods 1, 2 and 3
Population: All randomized participants who received at least 1 dose of study drug and had PSG measurements in Periods 1, 2 and 3.
Measure: Geometric Mean (90% Confidence Interval); unit: minutes (min)
Groups:
- 0.1 mg LY2624803: Single dose of 0.1 mg LY2624803 solution plus 1 placebo capsule administered orally in Periods 1, 2 and 3.
- 1.0 mg LY2624803: Single dose of one 1.0 mg LY2624803 capsule plus placebo solution administered orally in Periods 1, 2 and 3.
- 3.0 mg LY2624803: Single dose of one 3.0 mg LY2624803 capsule plus placebo solution administered orally in Periods 1, 2 and 3.
- 6.0 mg LY2624803: Single dose of one 6.0 mg LY2624803 capsule plus placebo solution administered orally in Periods 1, 2 and 3.
- Placebo: Single dose of 1 placebo capsule plus placebo solution administered orally in Periods 1, 2 and 3.
Arm/Group | 0.1 mg LY2624803 | 1.0 mg LY2624803 | 3.0 mg LY2624803 | 6.0 mg LY2624803 | Placebo
Number analyzed (Participants) | 8 | 17 | 16 | 8 | 17
minutes (min) | 58.88 [33.32 to 104.05] | 40.70 [25.67 to 64.54] | 32.27 [20.27 to 51.37] | 18.42 [10.44 to 32.51] | 61.10 [38.60 to 96.72]
Statistical Analysis 1: Comparison: 0.1 mg LY2624803 vs Placebo; Test type: Superiority or Other; p = 0.908, Mixed Models Analysis; Ratio of Geometric LS mean = 0.96, 90% CI 2-sided [0.56 to 1.65] — Ratio of Geometric LS mean is WASO of 0.1 mg LY2624803 / Placebo
Statistical Analysis 2: Comparison: 1.0 mg LY2624803 vs Placebo; Test type: Superiority or Other; p = 0.083, Mixed Models Analysis; Ratio of Geometric LS mean = 0.67, 90% CI 2-sided [0.45 to 0.98] — Ratio of Geometric LS mean is WASO of 1.0 mg LY2624803 / Placebo
Statistical Analysis 3: Comparison: 3.0 mg LY2624803 vs Placebo; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis; Ratio of Geometric LS mean = 0.53, 90% CI 2-sided [0.36 to 0.78] — Ratio of Geometric LS mean is WASO of 3.0 mg LY2624803 / Placebo
Statistical Analysis 4: Comparison: 6.0 mg LY2624803 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Ratio of Geometric LS mean = 0.30, 90% CI 2-sided [0.18 to 0.51] — Ratio of Geometric LS mean is WASO of 6.0 mg LY2624803 / Placebo

2. Secondary Outcome: Latency to Persistent Sleep (LPS)
Description: LPS is defined as the latency from the lights-off time to the first stage 2 sleep followed by at least 10 consecutive minutes of sleep epochs. Data presented are Geometric LS means. Geometric LS mean was calculated using mixed models analysis. The model included factors for treatment, treatment sequence, period and participants.
Time Frame: 8 hours in Periods 1, 2 and 3
Population: All randomized participants who received at least 1 dose of study drug and had PSG measurements in Periods 1, 2 and 3.
Measure: Geometric Mean (90% Confidence Interval); unit: min
Arm/Group | 0.1 mg LY2624803 | 1.0 mg LY2624803 | 3.0 mg LY2624803 | 6.0 mg LY2624803 | Placebo
Number analyzed (Participants) | 8 | 17 | 16 | 8 | 17
min | 14.30 [7.41 to 27.59] | 8.39 [5.41 to 13.02] | 7.84 [5.01 to 12.28] | 7.27 [3.78 to 13.99] | 10.40 [6.72 to 16.09]

3. Secondary Outcome: Total Sleep Time (TST)
Description: TST is defined as the total time in sleep epochs from sleep onset time to the end of the primary recording period (8 hours after lights -off). LS mean was calculated using mixed models analysis. The model included factors for treatment, treatment sequence, period and participants.
Time Frame: 8 hours in Periods 1, 2 and 3
Population: All randomized participants who received at least 1 dose of study drug and had PSG measurements in Periods 1, 2 and 3.
Measure: Least Squares Mean (90% Confidence Interval); unit: min
Arm/Group | 0.1 mg LY2624803 | 1.0 mg LY2624803 | 3.0 mg LY2624803 | 6.0 mg LY2624803 | Placebo
Number analyzed (Participants) | 8 | 17 | 16 | 8 | 17
min | 374.37 [333.21 to 415.53] | 404.35 [373.53 to 435.17] | 420.65 [389.43 to 451.88] | 452.09 [411.06 to 493.12] | 373.78 [343.12 to 404.44]

4. Secondary Outcome: PK: Maximum Plasma Concentration (Cmax) of LY2624803 After Single Oral Dose in Period 4
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 10, 12, 18, and 42 hours post-dose in Period 4
Population: All randomized participants who received a single oral dose of LY2624803 in Period 4 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- 0.1 mg LY2624803: Single dose of 0.1 mg LY2624803 solution plus 1 placebo capsule administered orally in Period 4
- 1.0 mg LY2624803: Single dose of one 1.0 mg LY2624803 capsule plus placebo solution administered orally in Period 4
- 3.0 mg LY2624803: Single dose of one 3.0 mg LY2624803 capsule plus placebo solution administered orally in Period 4
- 6.0 mg LY2624803: Single dose of one 6.0 mg LY2624803 capsule plus placebo solution administered orally in Period 4
Arm/Group | 0.1 mg LY2624803 | 1.0 mg LY2624803 | 3.0 mg LY2624803 | 6.0 mg LY2624803
Number analyzed (Participants) | 6 | 5 | 6 | 5
nanograms/milliliter (ng/mL) | 4.88 (10) | 43.8 (10) | 146 (13) | 251 (9)

5. Secondary Outcome: PK: Area Under the Concentration-Time Curve From Time 0 to Infinity [AUC(0-∞)] of LY2624803 After Single Oral Dose in Period 4
Time Frame: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 10, 12, 18, and 42 hours post-dose in Period 4
Population: All randomized participants who received a single oral dose of LY2624803 in Period 4 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms•hour/milliliter (ng•hr/mL)
Arm/Group | 0.1 mg LY2624803 | 1.0 mg LY2624803 | 3.0 mg LY2624803 | 6.0 mg LY2624803
Number analyzed (Participants) | 6 | 5 | 6 | 5
nanograms•hour/milliliter (ng•hr/mL) | 79.0 (39) | 714 (20) | 2240 (34) | 4220 (24)

ADVERSE EVENTS:
Groups:
- 0.1 mg LY2624803 - Periods 1-3: Single dose of 0.1 mg LY2624803 solution plus 1 placebo capsule administered orally in Periods 1, 2 and 3.
- 1.0 mg LY2624803 - Periods 1-3: Single dose of one 1.0 mg LY2624803 capsule plus placebo solution administered orally in Periods 1, 2 and 3.
- 3.0 mg LY2624803 - Periods 1-3: Single dose of one 3.0 mg LY2624803 capsule plus placebo solution administered orally in Periods 1, 2 and 3.
- 6.0 mg LY2624803 - Periods 1-3: Single dose of one 6.0 mg LY2624803 capsule plus placebo solution administered orally in Periods 1, 2 and 3.
- Placebo - Periods 1-3: Single dose of 1 placebo capsule plus placebo solution administered orally in Periods 1, 2 and 3.
- 0.1 mg LY2624803 - Period 4: Single dose of 0.1 mg LY2624803 solution plus 1 placebo capsule administered orally in Period 4.
- 1.0 mg LY2624803 - Period 4: Single dose of one 1.0 mg LY2624803 capsule plus placebo solution administered orally in Period 4.
- 3.0 mg LY2624803 - Period 4: Single dose of one 3.0 mg LY2624803 capsule plus placebo solution administered orally in Period 4.
- 6 mg LY2624803 - Period 4: Single dose of one 6.0 mg LY2624803 capsule plus placebo solution administered orally in Period 4.
Arm/Group | 0.1 mg LY2624803 - Periods 1-3 | 1.0 mg LY2624803 - Periods 1-3 | 3.0 mg LY2624803 - Periods 1-3 | 6.0 mg LY2624803 - Periods 1-3 | Placebo - Periods 1-3 | 0.1 mg LY2624803 - Period 4 | 1.0 mg LY2624803 - Period 4 | 3.0 mg LY2624803 - Period 4 | 6 mg LY2624803 - Period 4
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/17 | 0/17 | 0/8 | 0/18 | 0/6 | 0/5 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 2/9 | 3/17 | 3/17 | 0/8 | 3/18 | 0/6 | 2/5 | 1/6 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.1 mg LY2624803 - Periods 1-3 (N=9) | 1.0 mg LY2624803 - Periods 1-3 (N=17) | 3.0 mg LY2624803 - Periods 1-3 (N=17) | 6.0 mg LY2624803 - Periods 1-3 (N=8) | Placebo - Periods 1-3 (N=18) | 0.1 mg LY2624803 - Period 4 (N=6) | 1.0 mg LY2624803 - Period 4 (N=5) | 3.0 mg LY2624803 - Period 4 (N=6) | 6 mg LY2624803 - Period 4 (N=5)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days